CLINICAL TRIAL: NCT06354686
Title: Characterizing the Scalp Tolerability of Transcranial Magnetic Stimulation by Location and Stimulation Parameters
Brief Title: Characterizing the Scalp Tolerability of TMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Kevin A. Johnson, PhD RN, Research Faculty, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00004245
Record Dates: First submitted 2023-07-31; First posted 2024-04-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): This will be a single arm study with measurements of scalp location and TMS stimulation parameters.
  Interventions: Device: TMS Tolerability

INTERVENTIONS:
Device: TMS Tolerability — The primary objective is to characterize the tolerability of TMS by scalp location (over parietal, motor, modified Beam F3 prefrontal, THREE-D prefrontal, orbitofrontal, and medial prefrontal) and stimulation parameters (single pulse, 10 Hz, theta burst). The secondary objective is to evaluate the feasibility of the knee as a surrogate location to safely trial TMS parameters.

SUMMARY:
The primary objective is to characterize the tolerability of TMS by scalp location (over parietal, motor, modified Beam F3 prefrontal, THREE-D prefrontal, orbitofrontal, and medial prefrontal) and stimulation parameters (single pulse, 10 Hz, theta burst). The secondary objective is to evaluate the knee as a surrogate location to safely trial tolerability of novel TMS parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 years and older.
2. Capable to give informed written consent, ability to understand study procedures, and ability to comply with procedures for the entire length of the study.
3. Individuals with and without prior exposure to TMS are eligible (including individuals who have received TMS to treat depression).

Exclusion Criteria:

1. Medical contraindication for neuromodulation (e.g., ferrous metal in head, seizure disorder, brain tumor, stroke, aneurysm, multiple sclerosis, etc.).
2. Contraindication for scalp sensitivity and tolerability testing (e.g., sunburn, active headache, history of frequent and severe headaches).
3. Contraindication for knee sensitivity and tolerability testing (e.g., current knee injury or ongoing complications from prior history of knee surgery), unless knee testing skipped at the investigators' discretion.
4. Contraindication for participants with metal in both knees, unless knee testing skipped at the investigators' discretion.
5. Active substance use disorder in last 3 months or any current substance use that puts the participant at increased risk or significant impairment
6. Dementia or other cognitive disorder making unable to engage in study.
7. Any history or diagnosis of Schizophrenia, Schizoaffective Disorder, Delusional Disorder or other psychotic illness.
8. Taking any medication that significantly lowers the seizure threshold (e.g., tricyclic antidepressants, clozapine, etc.).
9. Any medication or substance use that significantly impacts sensory and tolerability measures based on the investigators' review of dosing and effect (e.g., topical anesthetics, botulinum toxin injections, ketamine, NSAIDS, opioids, anticonvulsants used in pain management, etc.).
10. Current, planned, or suspected pregnancy.
11. Unstable medical conditions or any current medical condition that could preclude being able to safely participate in TMS treatment (e.g., unstable metabolic abnormality, unstable angina, etc.).
12. Significant ongoing litigation or claims that impact research activities, as determined by the research study team. (Research may especially be impacted when mental health or pain is being evaluated for litigation or claims, such as civil and criminal cases, disability claims and worker's compensation).

The investigators will exclude the following individuals:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Tolerability of TMS - Scalp Location | 3-36 months
  Characterization of the tolerability of TMS by scalp location (over parietal, motor, modified Beam F3 prefrontal, THREE-D prefrontal, orbitofrontal, and medial prefrontal) using the McGill Pain Questionnaire and;
Tolerability of TMS - Stimulation parameters (single pulse, 10 Hz, theta burst). | 3-36 months
  Characterization of the tolerability of TMS by stimulation parameters (single pulse, 10 Hz, theta burst) using the McGill Pain Questionnaire.

SECONDARY OUTCOMES:
Tolerability of TMS (Knee Location) | 3-36 months
  Evaluation of the knee as a surrogate location to safely trial tolerability of TMS parameters. Qualitative descriptors (McGill Pain Questionnaire) will be selected by participants from a list of words and used to describe the quality of the TMS pulse (e.g. flickering, pricking, sharp, pinching, tugging, tingling, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No